CLINICAL TRIAL: NCT03589729
Title: Cardioprotection With Dexrazoxane in Acute Myeloid Leukemia (AML), High-Risk Myelodysplastic Syndrome (MDS), Myeloid Blast Phase of Chronic Myeloid Leukemia (CML), Ph+ AML, and Myeloid Blast Phase of Myeloproliferative Neoplasms
Brief Title: Dexrazoxane Hydrochloride in Preventing Heart-Related Side Effects of Chemotherapy in Participants With Blood Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0937; NCI-2018-01108 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0937 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-07-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Blasts 10 Percent or More of Bone Marrow Nucleated Cells; High Risk Myelodysplastic Syndrome; Myeloid Sarcoma; Myeloproliferative Neoplasm; Philadelphia Chromosome Positive
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Blast Crisis; Sarcoma, Myeloid; Myeloproliferative Disorders | interventions — Cladribine; Cytarabine; Dexrazoxane; Razoxane; Gemtuzumab; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (dexrazoxane hydrochloride, chemotherapy) (Experimental): See detailed description.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Dexrazoxane Hydrochloride; Drug: Gemtuzumab Ozogamicin; Drug: Idarubicin

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexrazoxane Hydrochloride — Given IV
  Other Names: Cardioxane; Totect; Zinecard
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR

SUMMARY:
This phase II trial studies how well dexrazoxane hydrochloride works in preventing heart-related side effects of chemotherapy in participants with blood cancers, such as acute myeloid leukemia, myelodysplastic syndrome, chronic myeloid leukemia, and myeloproliferative neoplasms. Chemoprotective drugs, such as dexrazoxane hydrochloride, may protect the heart from the side effects of drugs used in chemotherapy, such as cladribine, idarubicin, cytarabine, and gemtuzumab ozogamicin, in participants with blood cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the percentage of patients experiencing a decrease in left ventricular ejection fraction (LVEF) of 10 percent from baseline or decrease in LVEF below the normal limit of 50% during treatment with dexrazoxane (dexrazoxane hydrochloride) combined with cladribine, idarubicin, cytarabine, and Mylotarg (gemtuzumab ozogamicin) within the first 6-months of treatment.

SECONDARY OBJECTIVES:

I. To estimate the incidence of these cardiac symptoms while on dexrazoxane combined with idarubicin-based treatment: clinical heart failure, exertional dyspnea, orthopnea, S3 gallop, acute coronary syndrome, acute pulmonary edema and life-threatening arrhythmias.

II. To assess and monitor the change of troponin I (while still standard of care at MD Anderson) and high-sensitivity troponin T during treatment.

III. Collect safety/toxicity profile. IV. To assess rates of complete remission (CR)/complete remission with incomplete blood count recovery (CRi). (Cohorts 1-3) V. Other efficacy endpoints of interest include overall response, overall survival, event-free survival and remission duration. (Cohorts 1-3) VI. To assess the recurrence-free survival rate at 6 months. (Cohort 4)

EXPLORATORY OBJECTIVES:

I. To assess the metal chelation effects of dexrazoxane combined with chemotherapy (Mylotarg, cladribine, idarubicin, and cytarabine) by quantifying concentrations of toxic and essential metals and isotopic abundance ratios of blood and bone marrow before and during treatment.

II. To study and describe the relationship between pretreatment patient / disease characteristics (including cytogenetic and molecular abnormalities) and clinical outcomes.

III. To identify molecular biomarkers predictive of response to therapy. IV. To study and describe the relationship between patient / disease characteristics, use of intrathecal prophylaxis, and incidence of leptomeningeal disease.

V. To observe rates of fungal and other infections on the regimen. VI. To study environmental exposure data based on an environmental health assessment survey.

VII. To explore the impact of minimal residual disease (MRD) on relapse.

OUTLINE:

INDUCTION PHASE: Participants receive gemtuzumab ozogamicin intravenously (IV) over 2 hours on days 1, 4, and 7, cladribine IV over 1-2 hours on days 1-5, dexrazoxane hydrochloride IV over 15 minutes on days 1-3, idarubicin IV over 30 minutes on days 1-3, and cytarabine IV over 2 hours on days 1-5. Treatment repeats every 3-7 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION PHASE: After induction phase, participants receive gemtuzumab ozogamicin IV over 2 hours on day 1, cladribine IV over 1-2 hours on days 1-3, dexrazoxane hydrochloride IV over 15 minutes on days 1-2, idarubicin IV over 30 minutes on days 1-2, and cytarabine IV over 2 hours on days 1-3. Treatment repeats every 3-7 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Participants who go into remission or who are already in remission receive gemtuzumab ozogamicin IV over 2 hours on day 1 of course 1 and then every 2-3 months as needed. Participants also receive dexrazoxane hydrochloride IV over 15 minutes and idarubicin IV over 30 minutes on day 1, and cytarabine subcutaneously (SC) on days 1-7. Courses repeat every 3-7 weeks for 32 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Baseline left ventricular ejection fraction (LVEF) is greater than or equal to 50% by echocardiography (echo) or multigated acquisition (MUGA) scan.
* Patients of child bearing potential should use contraception.
* Patients with a diagnosis of acute myeloid leukemia (AML), or high risk myelodysplastic syndrome (MDS) (>= 10% blasts or International Prognostic Scoring System [IPSS] >= intermediate-2) or high-risk myeloproliferative neoplasm will be eligible.
* Patients with untreated or previously untreated chronic myeloid leukemia (CML) in myeloid blast phase or (Philadelphia chromosome-positive (Ph+) AML are also eligible.
* Patients with myeloproliferative neoplasms in blast phase will be eligible.
* Patients with isolated extramedullary myeloid neoplasm will be eligible.
* Patients with active CNS (central nervous system) disease are eligible.
* Bilirubin < 2mg/dL.
* AST (aspartate aminotransferase) and/or ALT (alanine aminotransferase) < 3 x ULN (upper limit of normal) - or < 5 x ULN if related to leukemic involvement.
* Creatinine < 1.5 x ULN.
* Hyperbilirubinemia is allowed if due to Gilbert's hyperbilirubinemia.
* A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
* Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.
* Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.
* Prior therapy for any of the cohorts may include with hydroxyurea, rescue doses of cytarabine, various combination-chemotherapy regimens, hematopoietic growth factors, azacytidine, decitabine, ATRA (all-trans retinoic acid).
* Cohort 1: Frontline cohort patients are eligible in the frontline cohort if they are untreated or previously treated already in CR if they received 3 or fewer cycles of previous chemotherapy (including either 1 induction and 2 consolidations or 2 inductions and 1 consolidation).
* Cohort 2: Salvage cohort in 1st and 2nd salvage patients are eligible in the salvage cohort 2 if they have active disease after first or second relapse or if they are in CR after previously documented first or second relapse as long as they if they have received 3 or fewer cycles of chemotherapy to achieve the most current CR.
* Cohort 3: Salvage cohort in 3rd salvage and beyond patients may be eligible in salvage cohort 3 if they have active disease after 3rd or greater relapse or if they are in CR after a previously documented relapse (3rd or greater), but may have only received 3 or fewer cycles of chemotherapy to achieve the most current CR.
* Cohort 4: Maintenance cohort: Patients in CR who are considered by treating physician to benefit from maintenance therapy are eligible for maintenance therapy with dexrazoxane combined with idarubicin plus cytarabine.

Exclusion Criteria:

* Any condition, including the presence of laboratory abnormalities, which judged by the investigator, places the patient at unacceptable risk.
* Active heart disease defined as: Unstable coronary syndromes, unstable or severe angina, recent myocardial infarction (MI) within 6 months.
* Decompensated heart failure (HF).
* Clinically significant arrhythmias.
* Severe valvular disease.
* History of coronary artery disease (CAD).
* Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
* Psychiatric illness/social situations that would limit compliance with study requirements per the judgment of the investigator.
* Patient with documented hypersensitivity to any of the components of the chemotherapy program.
* Men and women of childbearing potential who do not practice contraception.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients experiencing a decrease in left ventricular ejection fraction (LVEF) | Baseline up to 6 months
  Will assess a decrease in LVEF of 10 percent from baseline or decrease in LVEF below the normal limit of 50% during treatment with dexrazoxane hydrochloride combined with cladribine, idarubicin, cytarabine, and gemtuzumab ozogamicin.

SECONDARY OUTCOMES:
Incidence of cardiac symptoms | Up to 1 year
  Cardiac symptoms to be evaluated include: clinical heart failure, exertional dyspnea, orthopnea, S3 gallop, acute coronary syndrome, acute pulmonary edema and life-threatening arrhythmias
Assessment of change in troponin I and high-sensitivity troponin T | Up to 1 year
  Troponin levels will be collected before and after the day 1 dose of idarubicin each month during induction, consolidation, and maintenance therapy.
Incidence of adverse events | Up to 1 year
Complete remission (CR) /complete remission with incomplete blood count recovery (CRi) rates (Cohorts 1-3) | Up to 1 year
Overall response (Cohorts 1-3) | Up to 1 year
Overall survival (Cohorts 1-3) | Up to 1 year
Event-free survival (Cohorts 1-3) | Up to 1 year
Remission duration (Cohorts 1-3) | Up to 1 year
Recurrence-free survival | Up to 6 months
  The recurrence-free survival rate at 6 months will be a binary endpoint where the recurrence including death occurred within 6 months of treatment will be considered as "recurrence event".

OTHER OUTCOMES:
Assessment of metal chelation effects of dexrazoxane and chemotherapy | Up to 1 year
  Metal chelation effects assessed by utilizing technologies commonly used in the geochemistry.
Assessment of minimal residual disease (MRD) | Up to 1 year
  Will explore the impact of MRD on relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Maro Ohanian, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org